CLINICAL TRIAL: NCT01632904
Title: Polycythemia Vera Symptom Study Evaluating Ruxolitinib Versus Hydroxyurea in a Randomized, Multicenter, Double-Blind, Double-Dummy, Phase 3 Efficacy and Safety Study of Patient Reported Outcomes
Brief Title: Randomized Switch Study From Hydroxyurea to Ruxolitinib for RELIEF of Polycythemia Vera Symptoms: The Relief Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18424-357
Record Dates: First submitted 2012-06-29; First posted 2012-07-03 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Polycythemia Vera
Keywords: Polycythemia Vera; PV
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib; Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ruxolitinib and hydroxyurea (HU)-placebo (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: HU-placebo
- HU and ruxolitinib-placebo (Active Comparator)
  Interventions: Drug: Hydroxyurea (HU); Drug: Ruxolitinib-placebo

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib will be orally self-administered at a starting dose of 10 mg (two 5 mg tablets) twice a day. Dose increases of 5 mg (1 tablet) in twice-daily increments are permitted after 4 weeks and again after 8 weeks of therapy for subjects who meet prespecified criteria for inadequate efficacy.
  Arms: ruxolitinib and hydroxyurea (HU)-placebo
Drug: Hydroxyurea (HU) — Hydroxyurea (500 mg capsules) will be orally self-administered at the dose that the subject was receiving previously. The dose may be increased after 4 weeks and again after 8 weeks of therapy to optimize efficacy for subjects meeting prespecified criteria.
  Arms: HU and ruxolitinib-placebo
Drug: HU-placebo — All placebo will be self-administered, and dosing will be the same as with the blinded dose.
  When adjustments are made to the ruxolitinib dose, the dose of HU-placebo will be adjusted concurrently.
  Arms: ruxolitinib and hydroxyurea (HU)-placebo
Drug: Ruxolitinib-placebo — All placebo will be self-administered, and dosing will be the same as with the blinded dose.
  When adjustments are made to the HU dose, the dose of ruxolitinib-placebo will be adjusted concurrently.
  Arms: HU and ruxolitinib-placebo

SUMMARY:
The purpose of the RELIEF study is to compare symptoms in polycythemia vera (PV) subjects treated with ruxolitinib versus subjects treated with hydroxyurea (HU) as measured by the percent of subjects who achieve a clinically meaningful symptom improvement (ie, total symptom score reduction of ≥ 50% reduction) at Week 16 compared to Baseline. The study is also designed to demonstrate that these responses are durable with continued treatment.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter, double-blind, double-dummy, randomized study. Only subjects with PV who have received HU for at least 12 weeks, have been receiving a stable dose before screening, and still have symptoms related to PV will be enrolled.

Subjects will be randomized (1:1) to 1 of 2 treatment arms:

A: ruxolitinib and HU-placebo B: HU and ruxolitinib-placebo

Subjects randomized to either arm may be eligible to transition to open-label ruxolitinib after Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must currently be reporting symptoms while on a stable dose of HU monotherapy and be eligible to continue HU on study after randomization.
* Before screening, the subject must have been receiving HU for at least 12 weeks AND be receiving a stable dose.
* Subjects must meet baseline symptom criteria
* Subjects should meet at least 1 of the following criteria:

  * No more than 2 phlebotomies within the 6 months before screening OR
  * No palpable splenomegaly.
* Subjects must have a hematocrit that can be controlled within 35% to 48% (inclusive) before randomization.

Exclusion Criteria:

* Subjects with inadequate liver or renal function at screening.
* Subjects with clinically significant infection that requires therapy
* Subjects with known active hepatitis A, B, or C at screening or with known HIV positivity.
* Subjects with an active malignancy over the previous 2 years
* Subjects with clinically significant cardiac disease (Class III or IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, M.D., Study Director — Incyte Corporation
Locations (70):
- United States (51):
  - Scottsdale, Arizona
  - Fayetteville, Arkansas
  - Burbank, California
  - Glendale, California
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - Aurora, Colorado
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Niles, Illinois
  - Springfield, Illinois
  - Ames, Iowa
  - Westwood, Kansas
  - Alexandria, Louisiana
  - Baltimore, Maryland
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Morristown, New Jersey
  - Somerville, New Jersey
  - Albany, New York
  - Armonk, New York
  - Mineola, New York
  - New York, New York
  - Canton, Ohio
  - Bethlehem, Pennsylvania
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Amarillo, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Garland, Texas
  - Houston, Texas
  - Longview, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Tyler, Texas
  - Salt Lake City, Utah
  - Alexandria, Virginia
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Belgium (2):
  - Antwerp
  - Bruges
- Germany (6):
  - Aachen
  - Berlin
  - Freiburg im Breisgau
  - Hamburg
  - Stuttgart
  - Ulm
- Galway, Ireland
- Italy (3):
  - Florence
  - Reggio Calabria
  - Varese
- Spain (3):
  - Barcelona
  - Pamplona
  - Salamanca
- United Kingdom (4):
  - Boston
  - Leicester
  - Nottingham
  - West Bromwich

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib: Ruxolitinib will be orally self-administered at a starting dose of 10 mg (two 5 mg tablets) twice a day. Dose increases of 5 mg (1 tablet) in twice-daily increments are permitted after 4 weeks and again after 8 weeks of therapy for subjects who meet prespecified criteria for inadequate efficacy.
  HU-placebo All placebo will be self-administered, and dosing will be the same as with the blinded dose.
  When adjustments are made to the ruxolitinib dose, the dose of HU-placebo will be adjusted concurrently.
- Hydroxyurea: Hydroxyurea (HU) (500 mg capsules) will be orally self-administered at the dose that the subject was receiving previously. The dose may be increased after 4 weeks and again after 8 weeks of therapy to optimize efficacy for subjects meeting prespecified criteria.
  Ruxolitinib-placebo All placebo will be self-administered, and dosing will be the same as with the blinded dose.
  When adjustments are made to the HU dose, the dose of ruxolitinib-placebo will be adjusted concurrently.
Period: Overall Study
Arm/Group | Ruxolitinib | Hydroxyurea
Started | 54 | 56
Completed | 47 (Patients still in the study as of data cutoff, 27MAR2014.) | 50 (Patients still in the study as of 27MAR2014, including those who crossed over to ruxolitinib)
Not Completed | 7 | 6
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Subject decision | 3 | 2
Not completed — Disease Progression | 0 | 1
Not completed — Reason for discontinuation not available | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Hydroxyurea | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.68) | 64.2 (12.68) | 63.7 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 22 | 52
  Male | 24 | 34 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 53 | 56 | 109
  Asian | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving a ≥ 50% Improvement From Baseline in Total Symptom Score-Cytokine (TSS-C) at Week 16, as Measured by the Modified Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) Diary
Description: Symptoms of polycythemia vera were assessed using a modified Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) electronic diary. Using the diary, patients rated the following symptoms on a scale from 0 (absent) to 10 (worst imaginable): tiredness, itching, muscle aches, night sweats, and sweats while awake. The total symptom score ranged from 0-50 and was calculated as the sum of the 5 symptom scores. A higher score indicates worse symptoms.
Time Frame: From Baseline to Week 16
Population: Intent-to-Treat (ITT); all subjects randomized in the study. For the overall TSS-C score, only those subjects with a baseline score of 0 and a Week 16 score of 0 or missing were excluded from the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib | Hydroxyurea
Number analyzed (Participants) | 53 | 54
Percentage of participants | 43.4 | 29.6
Statistical Analysis 1: Comparison: Ruxolitinib vs Hydroxyurea; Test type: Superiority or Other; p = 0.139, Chi-squared; Odds Ratio (OR) = 1.82, 95% CI 2-sided [0.82 to 4.04]

2. Secondary Outcome: Percentage of Subjects Achieving ≥ 50% Improvement From Baseline in the Individual Symptom Scores for TSS-C at Week 16
Description: The TSS-C cluster includes tiredness, itching, muscle aches, night sweats, and sweats while awake.
Time Frame: From Baseline to Week 16
Population: Intent-to-Treat (ITT); all subjects randomized in the study. For individual symptom scores within the TSS-C cluster, only those subjects with a baseline score of 0 and a Week 16 score of 0 or missing were excluded from the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib | Hydroxyurea
Number analyzed (Participants) | 53 | 54
Percentage of participants
  Tiredness (n= 50, 53) | 40.0 | 26.4
  Itching (n= 48, 50) | 54.2 | 32.0
  Muscle aches (n= 47, 49) | 38.3 | 30.6
  Night sweats (n= 42, 48) | 47.6 | 41.7
  Sweats while awake (n= 42, 46) | 54.8 | 34.8

3. Secondary Outcome: Proportion of Subjects Randomized to Ruxolitinib Who Achieved ≥ 50% Improvement From Baseline in Total Symptom Score-Cytokine and the Individual Symptom Scores at Week 16 That Were Maintained at Week 48
Description: Durable Response on TSS-C/individual symptoms defined as a ≥ 50% reduction in TSS-C/individual symptoms at Week 16 that were maintained at Week 48
Time Frame: Week 48
Population: Intent-to-Treat (ITT); all subjects randomized to Ruxolitinib in the study. For TSS-C/individual symptoms, subject without baseline value was excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 54
percentage of participants
  TSS-C | 31.5 [19.5 to 45.6]
  Tiredness | 24.1 [13.5 to 37.6]
  Itching | 37.0 [24.3 to 51.3]
  Muscle aches | 20.4 [10.6 to 33.5]
  Night sweats | 29.6 [18.0 to 43.6]
  Sweats while awake | 37.0 [24.3 to 51.3]

ADVERSE EVENTS:
Time Frame: The duration of the study up to Week 16. This time frame defines the blinded, comparative phase of the study where the majority of patients remained on their original randomized assignment and exposure between ruxolitinib and hydroxyurea was similar.
Arm/Group | Ruxolitinib | Hydroxyurea
Serious Adverse Events (participants affected / at risk) | 5/54 | 4/56
Other Adverse Events (participants affected / at risk) | 50/54 | 45/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=54) | Hydroxyurea (N=56)
Angina unstable (Cardiac disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Cerebral ischemia (Nervous system disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hemoglobin decreased (Investigations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=54) | Hydroxyurea (N=56)
Headache (Nervous system disorders) | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Fatigue (General disorders) | 11 | 6
Anemia (Blood and lymphatic system disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 6 | 3
Urinary tract infection (Infections and infestations) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Vision blurred (Eye disorders) | 3 | 0
Weight increased (Investigations) | 3 | 0
Dizziness (Nervous system disorders) | 7 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 1
Edema peripheral (General disorders) | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Disturbance in attention (Psychiatric disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Palpitations (Cardiac disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Paresthesia (Nervous system disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3
Bronchitis (Infections and infestations) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 2
Hypertension (Vascular disorders) | 2 | 4
Depression (Psychiatric disorders) | 1 | 3
Gout (Metabolism and nutrition disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 0 | 2
Constipation (Gastrointestinal disorders) | 4 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Platelet count decreased (Investigations) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 11
Chest pain (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.